CLINICAL TRIAL: NCT06715826
Title: Development and Clinical Translation of immunoPET Imaging Probes for Breast Cancer
Brief Title: Target-specific immunoPET Imaging of Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2024-095-A
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancer Metastatic
Keywords: Trop2; HER2; Breast Cancer; ImmunoPET
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trop2/HER2-targeted immunoPET imaging (Experimental): Enrolled patients will undergo a Trop2/HER2-targeted immunoPET/CT scanning.
  Interventions: Drug: [18F]F-RESCA-RT4; Drug: [18F]F-RESCA-RB14

INTERVENTIONS:
Drug: [18F]F-RESCA-RT4 — Enrolled patients will receive 0.05-0.1mCi/kg of [18F]F-RESCA-RT4. ImmunoPET/CT imaging will be acquired 1 hour after [18F]F-RESCA-RT4 injection.
  Other Names: [18F]F-RT4
Drug: [18F]F-RESCA-RB14 — Enrolled patients will receive 0.05-0.1mCi/kg of [18F]F-RESCA-RB14. ImmunoPET/CT imaging will be acquired 1 hour after [18F]F-RESCA-RB14 injection.
  Other Names: [18F]F-RB14

SUMMARY:
The aim of this study is to establish and optimize the Trop2/HER2-targeted PET/CT imaging method, and its physiological and pathological distribution characteristics, on the basis of which the diagnostic efficacy of the above imaging agents in breast cancer will be evaluated.

DETAILED DESCRIPTION:
Enrolled patients will undergo whole-body[18F]F-RESCA-RT4(Trop2-targeted imaging probes ) or [18F]F-RESCA-RB14(HER2-targeted imaging probes) PET/CT scans at 1 hours after tracer injection(0.05-0.1 mCi/kg). Uptake of above imaging agents in tumor and normal organs/tissues will be scored visually and quantitatively.

Tumor uptake will be quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy will be calculated to evaluate the diagnostic efficacy. The correlation between lesion uptake and protein expression level determined by immunohistochemistry staining will be further analyzed. The exploration endpoint will be the imaging feasibility and preliminary diagnostic value of the above tracers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old and of female gender；
2. Histologically confirmed diagnosis of breast cancer or suspected breast cancer by diagnostic imaging;
3. Capable of giving signed informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol.

Exclusion Criteria:

1. Pregnancy；
2. Severe hepatic and renal insufficiency;
3. History of serious surgery in the last month;
4. Allergic to antibody or single-domain antibody radiopharmaceuticals.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2024-09-21 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of [18F]F-RESCA-RT4/ [18F]F-RESCA-RB14 | 1 day from injection of the tracer
  Measurement of the overall biodistribution of above probes in normal tissues and organs.
Standardized uptake value (SUV) | 1 day from injection of the tracer
  Standardized uptake value (SUV) of [18F]F-RESCA-RT4/ [18F]F-RESCA-RB14 in the included subjects' primary and/or metastatic lesions.
Radiation dosimetry of [18F]F-RESCA-RT4/[18F]F-RESCA-RB14 | 1 day from injection of the tracer
  Measurement of absorbed radiation doses (Gy/MBq) to tissues/organs, tumor(s), and whole body (Sv/MBq). Dynamic imaging within one hour will be acquired for the purpose.
The correlation between Trop2 expression and [18F]F-RESCA-RT4 uptake value | 60 days
  The Standardized uptake value (SUV) of [18F]F-RESCA-RT4 will be calculated, and the correlation between pathological results and tumor uptake of[18F]F-RESCA-T4 will be analyzed.
The correlation between HER2 expression and [18F]F-RESCA-RB14 uptake value | 60 days
  Standardized uptake value (SUV) of [18F]F-RESCA-RB14 will be calculated, and the correlation between pathological results and tumor uptake of [18F]F-RESCA-RB14 will be analyzed.
Diagnostic value of Trop2/HER2-targeted immunPET in patients with breast cancer | 30 days
  We will calculate the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and accuracy of [18F]F-RESCA-RT4/[18F]F-RESCA-RB14 PET/CT in patients with breast cancer. We will also compare the diagnostic value of above probes with that of traditional imaging tracers (e.g., 18F-FDG) and imaging modalities (e.g., MRI). All the above goals will be achieved by analyzing the static/dynamic[18F]F-RESCA-RT4/[18F]F-RESCA-RB14 PET/CT imaging data. Systematic evaluation of these parameters will elucidate the pharmacokinetics, pharmacodynamics, and, more importantly, the clinical value of [18F]F-RESCA-RT4/[18F]F-RESCA-RB14 PET/CT for patients with breast cancer.

SECONDARY OUTCOMES:
The predictive value of [18F]F-RESCA-RT4/ [18F]F-RESCA-RB14 in the course of targeted therapies | 3-6 months
  Baseline and follow-up [18F]F-RESCA-RT4/ [18F]F-RESCA-RB14 immunoPET imaging in targeted therapy will be investigated in this setting to determine the value of Trop2/HER2 immunoPET imaging in predicting or evaluating treatment responses.
Trop2/HER2-targeted immunPET in changing clinical decision-making for patients with breast cancer | 3-6 months
  After analyzing the imaging parameters and diagnostic/predictive value of [18F]F-RESCA-RT4/[18F]F-RESCA-RB14 PET/CT, we will also investigate how clinical use of [18F]F-RESCA-RT4/[18F]F-RESCA-RB14 PET/CT changes clinical decision-making for patients with breast cancer. Joint efforts from nuclear medicine physicians, breast surgeons, oncologists, and pathologists will draw solid conclusions from the imaging and clinical information.

CONTACTS AND LOCATIONS:
Overall Officials: Weijun Wei, Ph.D. & M.D., Study Chair — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China